CLINICAL TRIAL: NCT02819947
Title: Systemic Sclerosis Cohort in Seoul National University Hospital Single Center Prospective Cohort, of Patients With Systemic Sclerosis in Korea
Brief Title: Seoul National University Hospital Systemic Sclerosis Cohort
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Principal Investigator, Seoul National University Hospital
Other Study IDs: 2520140100
Record Dates: First submitted 2016-05-13; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; cohort; Korean
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: This is an observational prospective study. — Investigators will get clinical information including gender, date of birth, height, weight, family history for systemic sclerosis, education, and symptoms of organ involvement of skin, lung, heart, gastrointestinal tract, kidney, musculoskeletal system and laboratory data. Investigators will evaluate nailbed capillary microscope, hand x-ray, 6 minute walk test, echocardiography, computed tomography of chest, pulmonary function test (FVC%, DLCO%), and electrocardiogram as baseline. Investigators permit replacement of previous results within one year from baseline. Participants in the cohort will be followed up annually and investigators will treat SSc patients according to their routine practice in the best interest of patents. Medications for other comorbid conditions are allowed.

SUMMARY:
To establish a new prospective cohort of Korean patients with systemic sclerosis and track the natural history of the disease over time.

To generate new hypotheses for further investigation.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a multisystem and heterogeneous disease characterized by an unpredictable course and high morbidity and mortality. The complexity of SSc requires interdisciplinary diagnostic and therapeutic management and result in a growing burden for all health-care systems. For this reasons, researchers are seeking new diagnostic and therapeutic strategies to improve management of these patients. In order to improve clinical care and to develop recommendations for the diagnosis and treatment of SSc, disease registries are used to capture and track key patient information.

Therefore, SSc research associations and consortiums play a pivotal role to perform ongoing research and data collection to understanding the disease and support research projects. Currently, several national SSc registries in the UK, Germany, USA, Canada, Brazil, Australia and international registry, EUSTAR (European League Against Rheumatism scleroderma trial and research), have been established. However, the natural history of Asian populations are fully evaluated. Therefore, investigators decided to establish SSc cohort in Korean patients.

ELIGIBILITY:
Inclusion Criteria:

* SSc diagnosis according to 1980 or 2013 ACR classification criteria or 2001 criteria for the classification of early systemic sclerosis

Exclusion Criteria:

* When patients refuse to take part in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SSc diagnosis according to 1980 or 2013 ACR classification criteria or 2001 criteria for the classification of early systemic sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Internal organ involvement | 2-year
  Number of participants with internal organ involvement (Interstitial lung disease, Pulmonary arterial hypertension, Cardiac involvement, Gastrointestinal involvement, Renal involvement)

SECONDARY OUTCOMES:
Interstitial lung disease | 2-year
  Number of participants with ILD (at baseline and and during follow up) by computed tomography of chest
Interstitial lung disease-progression | 2-year
  Number of participants with progression of ILD from baseline by computed tomography of chest
Interstitial lung disease-Changes of FVC% from baseline | 2-year
  Changes of FVC% from baseline per year =FVC% at 1 year (0-unlimited%) - FVC% at baseline (0-unlimited%)
Interstitial lung disease-Changes of DLCO% from baseline | 2-year
  Changes of DLCO% from baseline per year =DLCO% at 1year (0-unlimited%) - DLCO% at baseline (0-unlimited%)
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Pulmonary arterial hypertension by echocardiography | 2-year
  Number of participants with pulmonary arterial hypertension (PAH) by electrocardiography
  -pulmonary arterial systolic pressure: 0-unlimited (mmHg)
Pulmonary arterial hypertension by right heart catheterization (optional) | 2-year
  Number of participants with PAH confirmed by right heart catheterization mean pulmonary arterial pressure: 0-unlimited (mmHg)
Abnormal cardiac function without other heart disease by echocardiography | 2-year
  Ejection fraction: 0-unlimited%
Pericardial effusion wihtout other heart disease by echocardiography | 2-year
  Pericardial effusion: mild, moderated, severe with hemodynamic unstability
Arrhythmia on electrocardiogram | 2-year
  Number of participants with arrhythmia on electrocardiogram
University of California Los Angeles Scleroderma Clinical Trials Consortium Gastrointestinal Scale (UCLA SCTC GIT) 2.0 | 2-year
  0-3 scale (0: no GI problems to 3: most severe)
Scleroderma-Specific Health Assessment Questionnaire (SHAQ) | 2-year
  0-3 (where 0 = without difficulty and 3 = unable to do)
Short Form(SF)-36 Health Survey | 2-year
  0-100 scale (a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability)

CONTACTS AND LOCATIONS:
Overall Officials: Eun Bong Lee, MD, PhD, Principal Investigator — Division of Rheumatology, Department of Internal Medicine, Seoul National University College of Medicine, Seoul, Korea
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gabrielli A, Avvedimento EV, Krieg T. Scleroderma. N Engl J Med. 2009 May 7;360(19):1989-2003. doi: 10.1056/NEJMra0806188. No abstract available. PMID 19420368
- [Result] Galluccio F, Walker UA, Nihtyanova S, Moinzadeh P, Hunzelmann N, Krieg T, Steen V, Baron M, Sampaio-Barros P, Kayser C, Nash P, Denton CP, Tyndall A, Muller-Ladner U, Matucci-Cerinic M. Registries in systemic sclerosis: a worldwide experience. Rheumatology (Oxford). 2011 Jan;50(1):60-8. doi: 10.1093/rheumatology/keq355. PMID 21148153